CLINICAL TRIAL: NCT06147440
Title: Different Dietary Patterns: Investigations in Healthy Participants
Brief Title: Different Dietary Patterns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ina Bergheim, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UVienna22
Record Dates: First submitted 2023-10-31; First posted 2023-11-27 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-04

CONDITIONS: Diet, Healthy; Endotoxemia
MeSH Terms: conditions — Endotoxemia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary pattern 1 (Experimental): Participants receive a standardized diet following the recommendation of DACH nutrition societies.
  Interventions: Other: Dietary intervention
- Dietary pattern 2 (Experimental): Participants receive a standardized diet following the recommendation of DACH nutrition societies.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Participants receive diets following different dietary patterns for 1 week.

SUMMARY:
The aim of the present study is to determine the effects of different standardized dietary patterns on general health markers, intestinal function, immune response and affective processes/ cognitive skills in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 kg/m² und 24.9 kg/m²

Exclusion Criteria:

* Chronic inflammatory diseases
* Metabolic diseases
* Viral or bacterial infections in the last 3 weeks
* Allergic reactions in the last 3 weeks
* Intake of anti-inflammatory drugs
* Malignant diseases
* Pregnancy and lactation
* Smoking
* Alcohol consumption > 10 g/d for women and > 20 g/d for men
* Drug consumption
* Vegetarian or vegan diet
* Food intolerances

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in parameters of intestinal barrier function | 1 week
  Changes in TLR ligand serum levels

SECONDARY OUTCOMES:
Changes in parameters of immune response | 1 week
  Changes in concentration of Interleukin-6 in cell culture supernatant of stimulated immune cells
Changes in blood lipid levels | 1 week
  Changes in triglyceride, cholesterol levels [mg/dl]
Changes in cognitive skills | 1 week
  Assessment of cognitive processes using computer-based psychological tasks (Stroop effect; calculation of differences in response times to incongruent vs. congruent word-color associations)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No